CLINICAL TRIAL: NCT01232660
Title: The Immunological Impact of Adding Hydroxychloroquine in Patients With Discordant CD4+ Cell Responses to Suppressive HAART: A Phase I Pilot Study.
Brief Title: Hydroxychloroquine for Discordant CD4 Responders on Highly Active Antiretroviral Therapy (HAART)
Acronym: SSAT039
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 039
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed (Active Comparator): Delayed addition of hydroxychloroquine in patients with discordant CD4+ cell responses to suppressive HAART
  Interventions: Drug: Hydroxychloroquine
- Immediate (Experimental): Immediate addition of hydroxychloroquine in patients with discordant CD4+ cell responses to suppressive HAART
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400mg once daily orally

SUMMARY:
The purpose of the study is to examine the effects of adding a drug called hydroxychloroquine, usually used to treat rheumatoid arthritis, to patients' usual antiretroviral combination. HIV causes activation of some parts of the immune system and this immune activation may persist despite effective antiretroviral therapy. Ongoing activation may be responsible for poor CD4 rise on antiretroviral therapy and for some HIV-related complications. Drugs like hydroxychloroquine work by inhibiting immune activation.

The study will primarily investigate the effect of adding this medication on immunological parameters (particularly CD4 count), on other safety parameters (such as cholesterol), patients' side effects and viral load.

If you decide to take part, the duration of your involvement in the study will be 24 weeks plus two screening visits up to 84 days prior to the start of the study and a follow up visit.

DETAILED DESCRIPTION:
Studies exploring changes in antiretrovirals or addition of antiretrovirals from new classes in patients with discordant immune response to suppressive HAART have, in general, yielded disappointing results.

The addition of the antiretroviral maraviroc (a CCR5 antagonist) in patients who had been on suppressive HAART for at least a year but with a CD4 count less than 250 (and not rising) yielded no improvement in CD4 counts in 6 individuals after approximately 5 months.

A small study investigating the benefit of switching to lopinavir/ritonavir (predominantly from NNRTI-based therapy) showed a significant improvement in CD4 cell count with a reduction in cell apoptosis at 6 months.However, data for other switches are lacking and lopinavir/ritonavir may not be a preferred switch option due to gastrointestinal tolerability and an increased risk of myocardial infarction in cohort analyses.

Chronic HIV infection is characterised by gradual loss of CD4 T-cells by direct (virus mediated CD4 death) and indirect mechanisms. Increased immune activation is an indirect mechanism that is central to CD4 T-cell loss. In observational studies, the level of immune activation is associated with the rate of CD4 decline and in patients taking antiretroviral therapy (with or without complete viral suppression) the extent of CD4 recovery is associated with the degree of immune activation.

Immune activation has also been shown to correlate with disease progression and survival. The causes of generalized immune activation in HIV are not fully understood but may be related to nef or gp120.

Hydroxychloroquine [Plaquanil®] is licensed to treat rheumatoid arthritis and other inflammatory conditions; it is related to the antimalarial chloroquine.

Hydroxychloroquine and chloroquine have long been used as immunomodulatory therapies for T-cell mediated disorders. The exact mechanisms of hydroxychloroquine are not fully understood, but the agent appears to affect T-cell proliferation and signalling. Hydroxychloroquine also inhibits T-cell proliferative responses and production of pro-inflammatory cytokines IL-1 and IL-6.

Hydroxychloroquine and chloroquine have been shown to inhibit HIV replication, regardless of viral clade or co-receptor tropism, and promote CD4 immune protection.

Three small clinical trials of hydroxychloroquine have been reported in HIV-infected patients. Hydroxychloroquine was associated with small to modest reductions in viral load both as monotherapy and as part of combination therapy. In one of these studies, hydroxychloroquine was compared with zidovudine in HIV-infected patients and patients in both groups had reduced levels of plasma HIV-1 RNA and serum p24 antigen after 16 weeks. Interleukin-6 (an inflammatory cytokine associated with increased risk of mortality in cohort studies of HIV) levels were significantly reduced in the hydroxychloroquine group but not in the zidovudine group.

The usual minimum effective dose of hydroxychloroquine is 400mg once daily (administered as two 200mg film-coated tablets) administered orally. This is also the dose selected for an ongoing Medical Research Council study investigating the immune benefits of hydroxychloroquine in treatment-naive patients not needing to start antiretrovirals. Hydroxychloroquine is cumulative in action and requires several weeks to exert its beneficial effects; for rheumatic disease, treatment should be discontinued if there is no improvement by 6 months. On this basis we feel that 3 months is sufficient time to detect most improvement in immune activation and 6 months sufficient time to observe any benefits if they occur. The maximum recommended dose of hydroxychloroquine is 6.5mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Age 18 to 65 years.
* On stable antiretroviral therapy for at least 96 weeks
* CD4 count less than 350 on screening blood test and on one other test performed within 4 months prior to screening and less than 150 cell rise in CD4 count in last 3 years
* Expression of CD38 on CD8+ T cells >10%
* Plasma HIV RNA viral load less than 50 copies/ml on screening blood test and for at least 72 weeks prior to screening (blips defined as a single viral load >50 and <500 copies/ml preceded and followed by an undetectable result will be permitted)
* Willing and able to provide written informed consent
* Females of child-bearing potential will need to use effective contraception
* Satisfactory ophthalmological assessment including:

  * visual acuity
  * careful ophthalmoscopy
  * fundoscopy
  * central visual field testing with a red target
  * colour vision.

Exclusion Criteria:

* History of psoriasis, porphyria cutanea tarda, epilepsy, myasthenia gravis, myopathy, cardiac arrhythmias or glucose 6-phosphate dehydrogenase (G6PD) deficiency.
* Insulin-dependent or non-insulin-dependent diabetes mellitus.
* Chronic liver disease of any cause or alcoholism (investigator defined)
* Pneumonia, meningitis, septicaemia or any other serious infection in the 2 months prior to screening.
* Any acute infection with fever and systemic symptoms in the last 24 hours.
* Any vaccinations in the 2 months prior to screening.
* Active malignancy (patients are eligible if treatment for the malignancy was completed more than 2 years prior to screening and there has been no subsequent clinical evidence of active disease or localised completely excised cutaneous cancers and low volume Kaposi's sarcoma) or any active immune-mediated or inflammatory disease.
* Any known suicide attempts (at any time in the past) or current or past history of depression requiring treatment within the 2 years prior to screening.
* A woman who is currently pregnant or breastfeeding.
* Use of systemic corticosteroids or other immunomodulatory drugs within the 12 months prior to screening.
* Current use of medication with known serious hepatotoxic effects or known interaction with hydroxychloroquine (section 5.2)
* Evidence of cardiac conduction defects or cardiac arrhythmia on screening ECG.
* Hepatitis B surface antigen (HBsAg) positive or Hepatitis C PCR positive (patients who are Hepatitis C antibody positive are allowed to enter if PCR is negative).
* Any of the following laboratory abnormalities on screening blood test:

  * Haemoglobin less than 10.5g/dl
  * Absolute neutrophil count less than 1.0x109/L
  * Platelet count less than 100 X 109/L
  * ALT or AST, or alkaline phosphatase above 2.5 x upper limit of normal (ULN) Template V 2.0, 06 April 2008 SSAT039 Page 23 of 73 Version 6.0, 17 October 2011
  * Serum creatinine greater than 1.5xULN
  * Estimated creatinine clearance (MDRD equation*) below 60ml/min
* Inability to attend or comply with treatment or follow-up scheduling.
* Current participation in any other clinical intervention trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in CD4 from baseline | 12 weeks
  To measure the change in CD4 from baseline after 12 weeks of hydroxychloroquine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Laura Waters, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom